CLINICAL TRIAL: NCT03743415
Title: Improving Informal Caregivers' and Cancer Survivors' Psychological Distress, Symptom Management and Health Care Use
Brief Title: Caregivers' and Cancer Survivors' Psychological Distress & Symptom Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1804501501; R01CA224282 (NIH)
Record Dates: First submitted 2018-07-20; First posted 2018-11-16 (Actual); Results first posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Cancer
Keywords: psychosocial oncology; symptom management
MeSH Terms: conditions — Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: This project will determine which dyads require which intervention sequence: Handbook alone, Handbook alone stepped up with Telephone Interpersonal Counseling (TIP-C) based on demonstrated needs after giving Handbook alone 4 weeks of time, or an combined TIP-C+Handbook for the first 8 weeks then Handbook alone for 4 weeks. Dyads will be initially randomized to either Handbook alone or TIP-C+Handbook. If the survivor's depression or anxiety does not respond to Handbook alone at week 4, dyads will be re-randomized to the TIPC+Handbook or continue with Handbook alone. Outcome data will be collected at baseline, weeks 13 (post-intervention) and 17 (follow-up). Total duration is 17 weeks.
Who Masked: Outcomes Assessor
Masking Description: Follow-up data collectors will be blind to the arm of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Handbook (Experimental): The Symptom Management and Survivorship Handbook is a self-care management handbook with each symptom chapter presented in an identical format: what the symptom is, how people describe the symptom, the causes of the symptom, strategies for managing the symptom and resources. The Handbook is available in English and Spanish. Each weekly call will begin with the symptom assessment. For each symptom rated at 4 or higher on a 0-10 scale of severity, the survivors will be referred for symptom self-management. During weeks 2-12, Handbook use since the last call (intervention enactment) and symptoms will be assessed. During weekly calls to caregivers, the caregivers will be notified of symptoms above threshold experienced by survivors and directed to the Handbook. During weeks 2-12, Handbook use and symptoms are assessed, a summary of survivors' symptoms provided. Calls will last about 10 minutes.
  Interventions: Behavioral: Handbook
- TIP-C plus Handbook (Experimental): Each survivor and caregiver will receive one 40-minute telephone call per week for 12 weeks. The Telephone Interpersonal Counseling (TIP-C) intervention 8-week protocol is the same for both survivor and caregiver. During weekly contacts, the counselors target social support behaviors using interpersonal communications techniques. Counselors can personalize the counseling intervention for the specific needs or interests as expressed during sessions while still adhering to a structured protocol. The final 4 weeks will be Handbook only.
  Interventions: Behavioral: TIP-C plus Handbook

INTERVENTIONS:
Behavioral: Handbook — see arm/group descriptions
  Other Names: Symptom Management and Survivorship Handbook
  Arms: Handbook
Behavioral: TIP-C plus Handbook — see arm/group descriptions
  Other Names: Telephone Interpersonal Counseling plus Handbook
  Arms: TIP-C plus Handbook

SUMMARY:
Sample: The sample will be 298 ethnically diverse (30% Hispanic) survivors who have a new diagnosis or localized recurrence of solid tumor cancer and elevated depression or anxiety and their informal caregivers. Design: The investigators selected the SMART design for this study over alternative designs (e.g.,implementation designs) because the SMART design allows a precision or personalized approach to determine the right treatment at the right dose with the right sequence for the right survivor-caregiver dyad. SMART designs, although newer, show promise in developing the sequences of evidence-based interventions for more efficient and individualized patient- and caregiver-centered care. The investigators will use findings from this study to create an algorithm for clinically meaningful decision making about symptom management for survivors and their caregivers to be tested in future implementation/dissemination studies. The dyad (survivor-caregiver) will be randomly assigned to either: 1) Symptom Management and Survivorship Guideline (Handbook) alone or 2) Telephone Interpersonal Counseling (TIP-C) +Handbook for 8 weeks followed by continued Handbook alone for 4 weeks. During 12 weeks following initial randomization, all participants will receive weekly telephone contacts to assess symptoms, deliver the assigned intervention and assess its enactment and fidelity. After the initial 4 weeks in the Handbook alone group, the survivor's response to the intervention will be determined. If the survivor responds (defined as a reduced score on depression and/or anxiety), the dyad will continue with the Handbook alone for 8 more weeks. If the survivor is a non-responder (defined as no improvement or a worsening score for depression and/or anxiety), the dyad will be re-randomized to either continue with Handbook alone for 8 more weeks, or add 8 weeks of TIP-C. Outcomes will be assessed at baseline, weeks 13 and 17 for both members of the dyad.

DETAILED DESCRIPTION:
Informal caregivers, typically family members or friends, provide more than half of the care needed for the 5.7 million cancer survivors (defined as individuals from diagnosis to end-of-life) in the United States, often with negative consequences to their health. Caregivers assist with the management of the survivor's symptoms such as fatigue, pain and insomnia, and others.Psychological distress (depression and anxiety) has been reported in at least 30% of survivors and their caregivers who are not always prepared for the task of symptom management. This research assists both the caregiver and survivor (the dyad in this study) to manage the survivor's cancer- and treatment-related symptoms and the distress of both members of the dyad in a sample of 298 survivors with elevated depression or anxiety and their 298 caregivers. Dyads will be recruited during the survivor's chemotherapy or targeted therapy for a solid tumor, a time when symptom burden and psychological distress are particularly high.

The investigators will use two evidence-based interventions extensively tested against active and passive controls in traditional randomized controlled trials (RCTs). While overall efficacy of these interventions has been established, individuals differ in their responses. When an intervention does not initially work, clinical logic is to either extend the timeframe or prescribe a different intervention. Yet, these alternatives are seldom tested and not evidence-based. The proposed project advances beyond a traditional RCT of testing fixed "one size fits all" interventions to the sequential multiple assignment randomized trial (SMART) design to build the evidence base for intervention sequencing that accounts for heterogeneity of responses.

The first intervention, a printed symptom management and survivorship handbook (Handbook) with strategies for self-management of symptoms common during chemotherapy will be given to both survivor and caregiver (the dyad). Handbook strategies, if successfully enacted, produce positive symptom responses for the survivor. However, psychological distress of the survivor or the caregiver may diminish the receipt and enactment of the Handbook strategies and also exacerbate the severity of other symptoms which, in turn, produces poor symptom responses. Research by this team has documented dyadic effects where survivors' psychosocial distress impacts that of the caregiver and vice versa. The survivor's and caregiver's distress exhibit similar trajectories. Therefore, the second intervention tested in sequencing is the 8-week telephone interpersonal counseling intervention (TIP-C) to manage psychological distress of the dyad.

The dyad (survivor-caregiver) will be randomly assigned to either: 1) Symptom Management and Survivorship Guideline (Handbook) alone or 2) Telephone Interpersonal Counseling (TIP-C) +Handbook for 8 weeks followed by continued Handbook alone for 4 weeks. During 12 weeks following initial randomization, all participants will receive weekly telephone contacts to assess symptoms, deliver the assigned intervention and assess its enactment and fidelity. After the initial 4 weeks in the Handbook alone group, the survivor's response to the intervention will be determined. If the survivor responds (defined as a reduced score on depression and/or anxiety), the dyad will continue with the Handbook alone for 8 more weeks. If the survivor is a non-responder (defined as no improvement or a worsening score for depression and/or anxiety), the dyad will be re-randomized to either continue with Handbook alone for 8 more weeks, or add 8 weeks of TIP-C. Outcomes will be assessed at baseline, weeks 13 and 17 for both members of the dyad.

The following specific aims will be tested.

1. Determine if dyads in the TIP-C+Handbook as compared to the Handbook alone group created by the first randomization will have: a) lower depression, anxiety, and summed severity of 13 other symptoms at weeks 1-12, 13, and 17 (primary outcomes); b) lower use of healthcare services (hospitalizations, urgent care or emergency department [ED] visits) during 17 weeks (secondary outcomes); c) greater self-efficacy, social support, and lower caregiver burden during weeks 13 and 17 (potential mediators).
2. Among non-responders to the Handbook alone after 4 weeks, determine if dyads in TIP-C+Handbook as compared to the Handbook alone group created by the second randomization will have better primary and secondary outcomes and potential mediators at weeks 5-12, 13, and 17.
3. Test the interdependence in survivors' and caregivers' primary and secondary outcomes.
4. Determine which characteristics of the dyad are associated with responses to the Handbook alone during weeks 1-4 and optimal outcomes for the dyad during weeks 1-12, 13 and 17 so as to determine tailoring variables for the decision rules of individualized sequencing of interventions in the future.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the survivors are: 1) age 18 or older; 2) undergoing chemotherapy, hormonal therapy, or targeted therapy for a solid tumor cancer; 3) able to perform basic activities of daily living; 4) cognitively oriented to time, place, and person (determined by recruiter); 5) reporting severity of >2 on depression or >4 on anxiety using a 0-10 standardized scale; 6) able to speak and understand English or Spanish; 7) access to a telephone and 8) has a caregiver who can be in any relationship role (e.g., spouse, sibling, parent, friend) who can participate with them.

Inclusion criteria for the caregivers are: 1) age 18 or older; 2) able to speak and understand English or Spanish; 3) access to a telephone; 4) not currently receiving counseling and/or psychotherapy; and 5) not currently treated for cancer.

Exclusion Criteria:

* Exclusion criteria are: 1) diagnosis of a psychotic disorder in the health record; 2) nursing home resident; 3) bedridden; 4) currently receiving counseling and/or psychotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 908 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terry Badger, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share the findings and data with other researchers, the public, and key stakeholders based on the principles that NIH has articulated regarding the sharing of study results and resources. The University of Arizona agrees that data sharing is essential for expedited translation of research results into knowledge, products, and procedures to improve health.
  Sharing of study results Manuscript based on results from the proposed study will be published in peer-reviewed journals. The investigators will select "open access" options for these manuscripts whenever possible.
  Data Sharing Data from this study will be available to other researchers under the following conditions: 1) appropriate human subjects protection is in place; 2) data have been de-identified; and 3) study investigators have publicly presented and published key findings. Data and safety monitoring plan is described under Human Subjects.
Supporting Information: Study Protocol, SAP
Time Frame: Anticipate later part of 2022
Access Criteria: Data from this study will be available to other researchers under the following conditions: 1) appropriate human subjects protection is in place; 2) data have been de-identified; and 3) study investigators have publicly presented and published key findings. Data and safety monitoring plan is described under Human Subjects.

REFERENCES:
- [Derived] Warner EL, Sikorskii A, Cunicelli N, Badger T, Segrin C, Morrill KE, Rainbow J. Employment Productivity and Cancer-Related Psychological Symptoms Among Adult Cancer Dyads. J Occup Environ Med. 2025 May 1;67(5):e294-e301. doi: 10.1097/JOM.0000000000003334. Epub 2025 Jan 30. PMID 39905918
- [Derived] Badger T, Segrin C, Crane TE, Chalasani P, Arslan W, Hadeed M, Given CW, Sikorskii A. A sequential multiple assignment randomized trial of symptom management for cancer survivors during treatment and their informal caregivers. Support Care Cancer. 2024 Jul 18;32(8):523. doi: 10.1007/s00520-024-08734-6. PMID 39023547
- [Derived] Badger T, Segrin C, Crane T, Morrill K, Sikorskii A. Social determinants of health, psychological distress, and caregiver burden among informal cancer caregivers of cancer survivors during treatment. J Psychosoc Oncol. 2024;42(3):333-350. doi: 10.1080/07347332.2023.2248486. Epub 2023 Aug 23. PMID 37609806

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the University of Arizona Cancer Center in Tucson and Phoenix, AZ, Valleywise Health, a federally qualified health center in Phoenix, AZ, and the community. Recruitment took place between January 16, 2019, and January 1, 2022. Research recruiters approached survivors at clinic visits, explained the study, and answered questions. Recruiters determined eligibility and followed protocol for consenting both the survivor and caregiver.
Pre-assignment Details: 908 (N= 451 survivors, N=457 caregivers) consented. 59 caregivers dropped before baseline. 398 dyads (survivor and caregiver) were interviewed at baseline. 24 dyads were not randomized due to the following: caregivers with no survivor interview (N=15), survivor ineligible (N=2), could not be reached (N=6), and other (N=1). 374 dyads were randomized into one of two groups: Symptom Management and Survivorship Handbook (SMSH) (N=277), and Telephone Interpersonal Counseling (TIP-C) + SMSH (N=97).
Groups:
- Survivors-SMSH Alone for 4 Weeks, Depression/Anxiety Responders Continued With SMSH Alone Weeks 5-12; Caregivers-SMSH Alone for 4 Weeks, Depression/Anxiety Responders Continued: The Symptom Management and Survivorship Handbook is a self-care management handbook with each symptom chapter presented in an identical format: what the symptom is, how people describe the symptom, the causes of the symptom, strategies for managing the symptom and resources. The Handbook was available in English and Spanish. Each weekly call began with a symptom assessment. For each symptom rated at 4 or higher on a 0-10 scale of severity, survivors and caregivers were referred for symptom self-management. After 4 weeks, depression or anxiety responders in the SMSH alone group continued with the SMSH alone for weeks 5-12. Depression or anxiety responders are survivors who started at severe at onset and ended at moderate or mild at a given time point (e.g., week 4), and survivors who started at moderate and ended at mild. At week 13, the survivor and caregiver were each called to complete the second assessment and at week 17 they were called to complete the third and final assessment.
- Survivors-SMSH Alone for 4 Weeks, Depression/Anxiety Non-responders Continued SMSH Alone Weeks 5-12; Caregivers-SMSH Alone for 4 Weeks, Depression/Anxiety Non-responders Continued SMSH Alone Weeks 5-12: The Symptom Management and Survivorship Handbook is a self-care management handbook with each symptom chapter presented in an identical format: what the symptom is, how people describe the symptom, the causes of the symptom, strategies for managing the symptom and resources. The Handbook was available in English and Spanish. Each weekly call began with a symptom assessment. For each symptom rated at 4 or higher on a 0-10 scale of severity, the survivors were referred for symptom self-management. After 4 weeks, depression or anxiety non-responders in the SMSH alone group were rerandomized (as a dyad) to either continue the SMSH alone for 8 weeks or add TIPC for 8 weeks. Depression or anxiety non-responders are survivors who do not respond to either or both depression or anxiety symptoms. Depression or anxiety responders started at severe at onset and ended at moderate or mild at a given time point (e.g., week 4), and survivors who started at moderate and ended at mild. At week 13, the survivor and caregiver were each called to complete the second assessment and at week 17 they were called to complete the third and final assessment.
- Survivors- SMSH Alone for 4 Weeks, Depression/Anxiety Non-responders Continued SMSH+TIPC Weeks 5-12; Caregivers- SMSH Alone for 4 Weeks, Depression/Anxiety Non-responders Continued SMSH+TIPC Weeks 5-12: The Symptom Management and Survivorship Handbook (SMSH) is a self-care management handbook with each symptom chapter presented in an identical format: what the symptom is, how people describe the symptom, the causes of the symptom, strategies for managing the symptom, and resources. The SMSH was available in English and Spanish. Each weekly call began with a symptom assessment. For each symptom rated at 4 or higher on a 0-10 scale of severity, dyads were referred for symptom self-management. After 4 weeks, depression or anxiety non-responders in the SMSH alone group were rerandomized (as a dyad) to either continue the SMSH alone for 8 weeks or add TIPC for 8 weeks. Depression or anxiety non-responders are survivors who do not respond to either or both depression or anxiety symptoms. Depression or anxiety responders started at severe at onset and ended at moderate or mild at week 4, and survivors who started at moderate and ended at mild. The Telephone Interpersonal Counseling (TIPC) 8-week protocol was the same for both survivor and caregiver. During weekly contact, counselors targeted social support behaviors using interpersonal communication techniques. Counselors personalized the counseling intervention for the specific needs or interests as expressed during sessions while still adhering to a structured protocol. At week 13, the survivor and caregiver were each called to complete the second assessment. At week 17 they were called to complete the final assessment.
- Survivors SMSH+TIPC During Weeks 1-8 Followed by SMSH Alone During Weeks 9-12; Caregivers SMSH+TIPC During Weeks 1-8 Followed by SMSH Alone During Weeks 9-12: The Symptom Management and Survivorship Handbook is a self-care management handbook with each symptom chapter presented in an identical format: what the symptom is, how people describe the symptom, the causes of the symptom, strategies for managing the symptom and resources. The Handbook was available in English and Spanish. Each weekly call began with a symptom assessment. For each symptom rated at 4 or higher on a 0-10 scale of severity, the survivors were referred for symptom self-management. In addition to the SMSH, each survivor and caregiver received one 40-minute telephone call per week for 12 weeks. The Telephone Interpersonal Counseling (TIP-C) intervention 8-week protocol was the same for both survivor and caregiver. During weekly contacts, the counselors targeted social support behaviors using interpersonal communications techniques. Counselors personalized the counseling intervention for the specific needs or interests as expressed during sessions while still adhering to a structured protocol. The final 4 weeks were Handbook only.
- Survivor Drop-outs From SMSH Alone Prior to Week 4; Caregiver Drop-outs From SMSH Alone Prior to Week 4: The Symptom Management and Survivorship Handbook is a self-care management handbook with each symptom chapter presented in an identical format: what the symptom is, how people describe the symptom, the causes of the symptom, strategies for managing the symptom, and resources. The Handbook was available in English and Spanish. Each weekly call began with a symptom assessment. For each symptom rated at 4 or higher on a 0-10 scale of severity, survivors and caregivers were referred for symptom self-management. These participants were lost to attrition prior to the week 4 assessment for response or non-response.
Period: Overall Study
Arm/Group | Survivors-SMSH Alone for 4 Weeks, Depression/Anxiety Responders Continued With SMSH Alone Weeks 5-12 | Survivors-SMSH Alone for 4 Weeks, Depression/Anxiety Non-responders Continued SMSH Alone Weeks 5-12 | Survivors- SMSH Alone for 4 Weeks, Depression/Anxiety Non-responders Continued SMSH+TIPC Weeks 5-12 | Survivors SMSH+TIPC During Weeks 1-8 Followed by SMSH Alone During Weeks 9-12 | Caregivers-SMSH Alone for 4 Weeks, Depression/Anxiety Responders Continued | Caregivers-SMSH Alone for 4 Weeks, Depression/Anxiety Non-responders Continued SMSH Alone Weeks 5-12 | Caregivers- SMSH Alone for 4 Weeks, Depression/Anxiety Non-responders Continued SMSH+TIPC Weeks 5-12 | Caregivers SMSH+TIPC During Weeks 1-8 Followed by SMSH Alone During Weeks 9-12 | Survivor Drop-outs From SMSH Alone Prior to Week 4 | Caregiver Drop-outs From SMSH Alone Prior to Week 4
Started | 166 | 44 | 44 | 97 | 166 | 44 | 44 | 97 | 23 | 23
Completed | 158 | 41 | 37 | 87 | 160 | 42 | 41 | 88 | 0 | 0
Not Completed | 8 | 3 | 7 | 10 | 6 | 2 | 3 | 9 | 23 | 23
Not completed — Death | 5 | 3 | 1 | 4 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 4 | 5 | 5 | 2 | 2 | 5 | 9 | 10
Not completed — Lost to Follow-up | 2 | 0 | 2 | 1 | 1 | 0 | 1 | 4 | 13 | 13

BASELINE CHARACTERISTICS:
Groups:
- Caregivers- SMSH Alone for 4 Weeks, Depression/Anxiety Responders Continued w/ SMSH Alone Weeks 5-12: The Symptom Management and Survivorship Handbook is a self-care management handbook with each symptom chapter presented in an identical format: what the symptom is, how people describe the symptom, the causes of the symptom, strategies for managing the symptom and resources. The Handbook was available in English and Spanish. Each weekly call began with a symptom assessment. For each symptom rated at 4 or higher on a 0-10 scale of severity, survivors and caregivers were referred for symptom self-management. After 4 weeks, depression or anxiety responders in the SMSH alone group continued with the SMSH alone for weeks 5-12. Depression or anxiety responders are survivors who started at severe at onset and ended at moderate or mild at a given time point (e.g., week 4), and survivors who started at moderate and ended at mild. At week 13, the survivor and caregiver were each called to complete the second assessment and at week 17 they were called to complete the third and final assessment.
- Caregivers-SMSH Alone for 4 Weeks, Depression/Anxiety Non-responders Continued SMSH+TIPC Weeks 5-12: The Symptom Management and Survivorship Handbook (SMSH) is a self-care management handbook with each symptom chapter presented in an identical format: what the symptom is, how people describe the symptom, the causes of the symptom, strategies for managing the symptom, and resources. The SMSH was available in English and Spanish. Each weekly call began with a symptom assessment. For each symptom rated at 4 or higher on a 0-10 scale of severity, dyads were referred for symptom self-management. After 4 weeks, depression or anxiety non-responders in the SMSH alone group were rerandomized (as a dyad) to either continue the SMSH alone for 8 weeks or add TIPC for 8 weeks. Depression or anxiety non-responders are survivors who do not respond to either or both depression or anxiety symptoms. Depression or anxiety responders started at severe at onset and ended at moderate or mild at week 4, and survivors who started at moderate and ended at mild. The Telephone Interpersonal Counseling (TIPC) 8-week protocol was the same for both survivor and caregiver. During weekly contact, counselors targeted social support behaviors using interpersonal communication techniques. Counselors personalized the counseling intervention for the specific needs or interests as expressed during sessions while still adhering to a structured protocol. At week 13, the survivor and caregiver were each called to complete the second assessment. At week 17 they were called to complete the final assessment.
- Caregivers- SMSH+ TIPC: The Symptom Management and Survivorship Handbook is a self-care management handbook with each symptom chapter presented in an identical format: what the symptom is, how people describe the symptom, the causes of the symptom, strategies for managing the symptom and resources. The Handbook was available in English and Spanish. Each weekly call began with a symptom assessment. For each symptom rated at 4 or higher on a 0-10 scale of severity, the survivors were referred for symptom self-management. In addition to the SMSH, each survivor and caregiver received one 40-minute telephone call per week for 12 weeks. The Telephone Interpersonal Counseling (TIP-C) intervention 8-week protocol was the same for both survivor and caregiver. During weekly contacts, the counselors targeted social support behaviors using interpersonal communications techniques. Counselors personalized the counseling intervention for the specific needs or interests as expressed during sessions while still adhering to a structured protocol. The final 4 weeks were Handbook only.
- Total: Total of all reporting groups
Arm/Group | Survivors-SMSH Alone for 4 Weeks, Depression/Anxiety Responders Continued With SMSH Alone Weeks 5-12 | Survivors-SMSH Alone for 4 Weeks, Depression/Anxiety Non-responders Continued SMSH Alone Weeks 5-12 | Survivors- SMSH Alone for 4 Weeks, Depression/Anxiety Non-responders Continued SMSH+TIPC Weeks 5-12 | Survivors SMSH+TIPC During Weeks 1-8 Followed by SMSH Alone During Weeks 9-12 | Caregivers- SMSH Alone for 4 Weeks, Depression/Anxiety Responders Continued w/ SMSH Alone Weeks 5-12 | Caregivers-SMSH Alone for 4 Weeks, Depression/Anxiety Non-responders Continued SMSH Alone Weeks 5-12 | Caregivers-SMSH Alone for 4 Weeks, Depression/Anxiety Non-responders Continued SMSH+TIPC Weeks 5-12 | Caregivers- SMSH+ TIPC | Survivor Drop-outs From SMSH Alone Prior to Week 4 | Caregiver Drop-outs From SMSH Alone Prior to Week 4 | Total
Number analyzed (Participants) | 166 | 44 | 44 | 97 | 166 | 44 | 44 | 97 | 23 | 23 | 748
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.48 (11.86) | 61.61 (12.28) | 59.09 (13.77) | 60.44 (12.47) | 53.98 (16.04) | 54.14 (15.56) | 56.25 (16.07) | 53.89 (3.46) | 60.08 (14.43) | 52.56 (16.52) | 57.06 (13.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 38 | 33 | 78 | 112 | 30 | 34 | 59 | 16 | 17 | 541
  Male | 42 | 6 | 11 | 19 | 54 | 14 | 10 | 38 | 7 | 6 | 207
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 71 | 17 | 13 | 42 | 78 | 17 | 16 | 43 | 10 | 11 | 318
  Not Hispanic or Latino | 95 | 27 | 30 | 55 | 88 | 27 | 28 | 53 | 13 | 12 | 428
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 0 | 1 | 4 | 11 | 2 | 2 | 3 | 3 | 2 | 37
  Asian | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 6
  Black or African American | 3 | 0 | 1 | 3 | 4 | 0 | 0 | 2 | 0 | 1 | 14
  White | 94 | 29 | 28 | 54 | 94 | 26 | 26 | 62 | 12 | 11 | 436
  More than one race | 8 | 3 | 3 | 6 | 11 | 1 | 1 | 3 | 0 | 0 | 36
  Unknown or Not Reported | 49 | 12 | 10 | 30 | 44 | 14 | 14 | 26 | 7 | 8 | 214
Symptom Severity [Mean (Standard Deviation); unit: units on a scale] — Symptoms were measured using the General Symptom Distress Scale (GSDS) assessment of 18 symptoms: fatigue, sleep difficulty, pain, headache, difficulty concentrating, lack of appetite, nausea, vomiting, constipation, diarrhea, numbness or tingling, skin rashes or sores, swelling, weakness, shortness of breath, cough, depression, and anxiety. Respondents indicated the severity of each symptom (0= not present, 10= worst possible). A summed symptom severity index for 16 symptoms other than depression and anxiety was derived. The potential range is 0-160, a higher score reflects a worse outcome.
  units on a scale | 34.67 (22.28) | 43.55 (23.51) | 48.02 (30.12) | 43.53 (22.92) | 19.73 (18.00) | 22.00 (18.47) | 19.39 (16.31) | 20.61 (17.51) | 51.17 (26.01) | 21.17 (23.37) | 30.43 (23.72)

OUTCOME MEASURES:

1. Primary Outcome: Symptom Severity Index- Comparison of Two Groups Created by First Randomization
Description: Symptoms were measured using the modified General Symptom Distress Scale (GSDS), a brief instrument that measures 18 common symptoms fatigue, sleep difficulties, pain, headache, difficulty concentrating, lack of appetite, nausea, vomiting, constipation, diarrhea, numbness or tingling, skin rashes or sores, swelling, weakness, shortness of breath, cough, depression, and anxiety. Respondents indicate severity of each symptom on the scale from 0=not present to 10=worst possible. A summed symptom severity index for 16 symptoms other than depression and anxiety was computed by adding severities of 16 symptoms at each weekly contact (weeks 1-12) and week 13 interview for the immediate effects. The summed symptom severity range is 0-160, a higher score reflects a worse outcome. Week 17 value of the index was analyzed to determine the sustained effects.
Time Frame: Weeks 1-13 and week 17
Population: Out of 374 dyads (survivors and caregivers), 277 were randomized initially to the SMSH alone, and 97 to SMSH+TIPC.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Survivors- SMSH Alone: The Symptom Management and Survivorship Handbook is a self-care management handbook with each symptom chapter presented in an identical format: what the symptom is, how people describe the symptom, the causes of the symptom, strategies for managing the symptom and resources. The Handbook was available in English and Spanish. Each weekly call began with a symptom assessment. For each symptom rated at 4 or higher on a 0-10 scale of severity, the survivors were referred for symptom self-management. During weeks 2-12, Handbook use since the last call (intervention enactment) and symptoms were assessed. During weekly calls to caregivers, the caregivers were notified of symptoms above the threshold experienced by survivors and directed to the Handbook. During weeks 2-12, Handbook use and symptoms were assessed, and a summary of survivors' symptoms was provided. Calls lasted about 10 minutes.
  Handbook: see arm/group descriptions
- Survivors- SMSH+ TIPC; Caregivers- SMSH+ TIPC: Each survivor and caregiver received one 40-minute telephone call per week for 12 weeks. The Telephone Interpersonal Counseling (TIP-C) intervention 8-week protocol was the same for both survivor and caregiver. During weekly contacts, the counselors targeted social support behaviors using interpersonal communications techniques. Counselors personalized the counseling intervention for the specific needs or interests as expressed during sessions while still adhering to a structured protocol. The final 4 weeks were Handbook only.
  TIP-C plus Handbook: see arm/group descriptions
- Caregivers- SMSH Alone: The Symptom Management and Survivorship Handbook is a self-care management handbook with each symptom chapter presented in an identical format: what the symptom is, how people describe the symptom, the causes of the symptom, strategies for managing the symptom and resources. The Handbook was available in English and Spanish. Each weekly call began with a symptom assessment. For each symptom rated at 4 or higher on a 0-10 scale of severity, the survivors were referred for symptom self-management. During weeks 2-12, Handbook use since the last call (intervention enactment) and symptoms were assessed. During weekly calls to caregivers, the caregivers were notified of symptoms above the threshold experienced by survivors and directed to the Handbook. During weeks 2-12, Handbook use and symptoms were assessed, and a summary of survivors' symptoms was provided. The calls lasted about 10 minutes.
Arm/Group | Survivors- SMSH Alone | Survivors- SMSH+ TIPC | Caregivers- SMSH Alone | Caregivers- SMSH+ TIPC
Number analyzed (Participants) | 277 | 97 | 277 | 97
units on a scale
  Average over weeks 1-13 | 26.28 (0.60) | 26.55 (0.98) | 12.02 (0.40) | 11.19 (0.65)
  Week 17 | 25.72 (1.07) | 26.30 (1.78) | 10.16 (0.74) | 9.04 (1.15)
Statistical Analysis 1: Comparison: Survivors- SMSH Alone vs Survivors- SMSH+ TIPC; The null hypothesis was that the means of two groups were equal. The alternative hypothesis was that the means of two groups were not equal. The adjusted effect size d=0.54 between the SMSH alone group and SMSH+TIPC group was detectable with power of .94 in two-sided tests at .05 level of significance; Test type: Superiority — The key parameter was the coefficient for the trial arm difference in linear mixed effects model that reflected average difference between arms over time (weeks 1-13); p = .81, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Linear mixed effects models were used for 13 repeated measures of the symptom index, adjusting for baseline value; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-2.50 to 1.96], Standard Error of Mean 1.16 — Mean of SMSH alone minus mean of SMSH+TIPC
Statistical Analysis 2: Comparison: Survivors- SMSH Alone vs Survivors- SMSH+ TIPC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at week 17 in linear mixed effects model; p = .78, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; The model included adjustment for baseline value of the symptom index; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-4.65 to 3.49], Standard Error of Mean 2.07 — Mean of SMSH alone minus SMSH+TIPC
Statistical Analysis 3: Comparison: Caregivers- SMSH Alone vs Caregivers- SMSH+ TIPC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference in linear mixed effects model that included reflected average difference between arms over time (weeks 1-13); p = .27, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome was adjusted for in the model; Mean Difference (Final Values) = 0.83, 95% CI 2-sided [-0.66 to 2.32], Standard Error of Mean 0.76 — Mean of SMSH minus SMSH+TIPC
Statistical Analysis 4: Comparison: Caregivers- SMSH Alone vs Caregivers- SMSH+ TIPC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at week 17 in linear mixed effects model; p = .19, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome was adjusted for in the model; Mean Difference (Final Values) = 1.76, 95% CI 2-sided [-0.88 to 4.39], Standard Error of Mean 1.35 — Mean of SMSH alone minus SMSH+TIPC

2. Primary Outcome: Symptom Severity Index- Comparison of Two Groups Created by Second Randomization
Description: Symptoms were measured using the modified General Symptom Distress Scale (GSDS), a brief instrument that measures 18 common symptoms fatigue, sleep difficulties, pain, headache, difficulty concentrating, lack of appetite, nausea, vomiting, constipation, diarrhea, numbness or tingling, skin rashes or sores, swelling, weakness, shortness of breath, cough, depression, and anxiety. Respondents indicate severity of each symptom on the scale from 0=not present to 10=worst possible. A summed symptom severity index for 16 symptoms other than depression and anxiety was computed by adding severities of 16 symptoms at each weekly contact (weeks 5-12) and week 13 interview for the immediate effects. The summed symptom severity range is 0-160, a higher score reflects a worse outcome. Week 17 value of the index was analyzed to determine the sustained effects.
Time Frame: Weeks 5-13 and week 17
Population: Survivors and caregivers randomized for the second time after survivor's non-response to the SMSH alone after 4 weeks.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Survivors- SMSH Alone | Survivors- SMSH+ TIPC | Caregivers- SMSH Alone | Caregivers- SMSH+ TIPC
Number analyzed (Participants) | 44 | 44 | 44 | 44
units on a scale
  Average over weeks 5-13 | 33.67 (1.73) | 34.14 (1.75) | 14.50 (1.36) | 12.53 (1.37)
  Week 17 | 37.84 (2.73) | 35.86 (2.82) | 15.22 (1.95) | 11.92 (1.96)
Statistical Analysis 1: Comparison: Survivors- SMSH Alone vs Survivors- SMSH+ TIPC; The null hypothesis was that the means of two groups were equal. The alternative hypothesis was that the means of two groups were not equal. . The adjusted effect size (Cohen's d=0.54) was used to power comparisons on the primary outcomes reported by groups from the second randomization. This analysis indicated that 60 per group would be required for power of .80 or greater in two-sided tests at α= 0.05; Test type: Superiority — The key parameter was the coefficient for the trial arm difference in linear mixed effects model that included reflected average difference between arms over weeks 5-13; p = .53, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome was adjusted for in the model; Mean Difference (Final Values) = 2.43, 95% CI 2-sided [-3.30 to 6.36], Standard Error of Mean 2.46 — Mean of SMSH alone minus SMSH+TIPC
Statistical Analysis 2: Comparison: Survivors- SMSH Alone vs Survivors- SMSH+ TIPC; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at week 17 in linear mixed effects model; p = .97, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome was adjusted for in the model; Mean Difference (Final Values) = 1.99, 95% CI 2-sided [-5.70 to 9.68], Standard Error of Mean 3.92 — Mean of SMSH alone minus SMSH+TIPC
Statistical Analysis 3: Comparison: Caregivers- SMSH Alone vs Caregivers- SMSH+ TIPC; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = .31, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome was adjusted for in the model; Mean Difference (Final Values) = 1.96, 95% CI 2-sided [-1.83 to 5.75], Standard Error of Mean 1.94 — Mean of SMSH alone minus SMSH+TIPC
Statistical Analysis 4: Comparison: Caregivers- SMSH Alone vs Caregivers- SMSH+ TIPC; The null hypothesis was that the means of two groups were equal. The alternative hypothesis was that the means of two groups were not equal. The adjusted effect size (Cohen's d=0.54) was used to power comparisons on the primary outcomes reported by groups from the second randomization. This analysis indicated that 60 per group would be required for power of .80 or greater in two-sided tests at α= 0.05; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at week 17 in linear mixed effects model; p = .61, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome was adjusted for in the model; Mean Difference (Net) = 3.30, 95% CI 2-sided [-2.13 to 8.74], Standard Error of Mean 2.77 — Mean of SMSH minus SMSH+TIPC

3. Secondary Outcome: Depressive Symptoms- Comparison of Two Groups Created by First Randomization
Description: Measured using Center for Epidemiological Studies- Depression (CES-D) 20-item scale. Potential score range is 0-60. Higher scores indicated worse outcome (higher depressive symptoms).
Time Frame: Week 13 and week 17
Population: Survivors and caregivers included in the first randomization
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Survivors- SMSH Alone | Survivors- SMSH+ TIPC | Caregivers- SMSH Alone | Caregivers- SMSH+ TIPC
Number analyzed (Participants) | 277 | 97 | 277 | 97
units on a scale
  Week 13 | 12.90 (0.59) | 13.78 (0.97) | 10.48 (0.49) | 10.44 (0.83)
  Week 17 | 13.60 (0.60) | 13.67 (0.98) | 9.94 (0.49) | 9.62 (0.82)
Statistical Analysis 1: Comparison: Survivors- SMSH Alone vs Survivors- SMSH+ TIPC; The null hypothesis was that the means of two groups were equal. The alternative hypothesis was that the means of two groups were not equal. Sample size was determined by the power calculation for the primary outcome; Test type: Superiority — Key parameter was the difference between arms at week 13; p = .44, Regression, Linear — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome was adjusted for in the model; Mean Difference (Final Values) = -0.99, 95% CI 2-sided [-3.12 to 1.35], Standard Error of Mean 1.14 — Mean of SMSH minus SMSH+TIPC
Statistical Analysis 2: Comparison: Survivors- SMSH Alone vs Survivors- SMSH+ TIPC; The key parameter was the coefficient for the trial arm difference at week 17 in linear mixed effects model; Test type: Superiority — The null hypothesis was that the means of two groups were equal. The alternative hypothesis was that the means of two groups were not equal. Sample size was determined by the power calculation for the primary outcome; p = .95, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome was adjusted for in the model; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-2.32 to 2.18], Standard Error of Mean 1.15 — Mean of SMSH minus SMSH+TIPC
Statistical Analysis 3: Comparison: Caregivers- SMSH Alone vs Caregivers- SMSH+ TIPC; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at week 13 in linear mixed effects model; p = .97, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome was adjusted for in the model; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-1.85 to 1.93], Standard Error of Mean 0.96 — Mean of SMSH minus SMSH+TIPC
Statistical Analysis 4: Comparison: Caregivers- SMSH Alone vs Caregivers- SMSH+ TIPC; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at week 17 in linear mixed effects model; p = .74, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome was adjusted for in the model; Mean Difference (Final Values) = 0.32, 95% CI 2-sided [-1.56 to 2.20], Standard Error of Mean 0.96 — Mean of SMSH minus SMSH+TIPC

4. Secondary Outcome: Depressive Symptoms- Comparison of Two Groups Created by Second Randomization
Description: as for outcome 3
Time Frame: Week 13 and week 17
Population: Survivors and caregivers randomized for the second time after survivor's non-response to the SMSH alone after 4 weeks.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Survivors- SMSH Alone | Survivors- SMSH+ TIPC | Caregivers- SMSH Alone | Caregivers- SMSH+ TIPC
Number analyzed (Participants) | 44 | 44 | 44 | 44
units on a scale
  Week 13 | 19.21 (1.57) | 19.17 (1.65) | 11.60 (1.29) | 13.60 (1.29)
  Week 17 | 20.34 (1.58) | 21.24 (1.67) | 12.67 (1.27) | 12.46 (1.29)
Statistical Analysis 1: Comparison: Survivors- SMSH Alone vs Survivors- SMSH+ TIPC; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at week 13 in linear mixed effects model; p = .98, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome was adjusted for in the model; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-4.49 to 4.58], Standard Error of Mean 2.31 — Mean of SMSH minus mean of SMSH+TIPC
Statistical Analysis 2: Comparison: Survivors- SMSH Alone vs Survivors- SMSH+ TIPC; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at week 17 in linear mixed effects model; p = .70, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome was adjusted for in the model; Mean Difference (Final Values) = -0.90, 95% CI 2-sided [-5.48 to 3.68], Standard Error of Mean 2.34 — Mean of SMSH minus SMSH+TIPC
Statistical Analysis 3: Comparison: Caregivers- SMSH Alone vs Caregivers- SMSH+ TIPC; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at week 13 in linear mixed effects model; p = .27, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome was adjusted for in the model; Mean Difference (Final Values) = -2.00, 95% CI 2-sided [-5.62 to 1.62], Standard Error of Mean 1.85 — Mean of SMSH minus SMSH+TIPC
Statistical Analysis 4: Comparison: Caregivers- SMSH Alone vs Caregivers- SMSH+ TIPC; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at week 17 in linear mixed effects model; p = .91, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome was adjusted for in the model; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-3.40 to 3.81], Standard Error of Mean 1.84 — Mean of SMSH minus SMSH+TIPC

5. Secondary Outcome: Anxiety Symptoms- Comparison of Two Groups Created by First Randomization
Description: Measured using Patient-Reported Outcomes Measurement Information System (PROMIS)-Anxiety 8a short form. Each question is rated on a five-point scale from 1=Never to 5=Always. The lowest possible raw score is 8; the highest possible raw score is 40. Raw scores are converted into t-scores with potential range of 37.1 to 83.1. Higher scores indicate greater anxiety. The mean of the US general population is 50 with standard deviation 10. Consensus-based but not data-based thresholds for scores in cancer populations are 50 for mildly symptomatic, 60 for moderately symptomatic, and 70 for severely symptomatic.
Time Frame: Week 13 and week 17
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Survivors- SMSH Alone | Survivors- SMSH+ TIPC | Caregivers- SMSH Alone | Caregivers- SMSH+ TIPC
Number analyzed (Participants) | 277 | 97 | 277 | 97
T-score
  Week 13 | 48.98 (0.54) | 50.86 (0.90) | 47.72 (0.50) | 47.58 (0.83)
  Week 17 | 49.11 (0.54) | 50.91 (0.90) | 47.58 (0.50) | 46.89 (0.82)
Statistical Analysis 1: Comparison: Survivors- SMSH Alone vs Survivors- SMSH+ TIPC; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at week 13 in linear mixed effects model; p = .06, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome was adjusted for in the model; Mean Difference (Final Values) = -1.93, 95% CI 2-sided [-3.98 to 0.19], Standard Error of Mean 1.06 — Mean of SMSH minus SMSH+TIPC
Statistical Analysis 2: Comparison: Survivors- SMSH Alone vs Survivors- SMSH+ TIPC; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at week 17 in linear mixed effects model; p = .09, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome was adjusted for in the model; Mean Difference (Final Values) = -1.78, 95% CI 2-sided [-3.81 to 0.11], Standard Error of Mean 1.00 — Mean of SMSH minus SMSH+TIPC
Statistical Analysis 3: Comparison: Caregivers- SMSH Alone vs Caregivers- SMSH+ TIPC; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at week 13 in linear mixed effects model; p = .89, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome was adjusted for in the model; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-1.77 to 2.04], Standard Error of Mean 0.97 — Mean of SMSH minus SMSH+TIPC
Statistical Analysis 4: Comparison: Caregivers- SMSH Alone vs Caregivers- SMSH+ TIPC; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at week 17 in linear mixed effects model; p = .47, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome was adjusted for in the model; Mean Difference (Final Values) = 0.96, 95% CI 2-sided [-1.20 to 2.58], Standard Error of Mean 0.96 — Mean of SMSH minus SMSH+TIPC

6. Secondary Outcome: Anxiety Symptoms- Comparison of Two Groups Created by Second Randomization
Description: as for outcome 5
Time Frame: Week 13 and week 17
Population: Survivors and caregivers randomized for the second time after survivor's non-response to the SMSH alone after 4 weeks.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Survivors- SMSH Alone | Survivors- SMSH+ TIPC | Caregivers- SMSH Alone | Caregivers- SMSH+ TIPC
Number analyzed (Participants) | 44 | 44 | 44 | 44
T-score
  Week 13 | 52.90 (1.32) | 54.31 (1.39) | 50.47 (1.31) | 49.92 (1.30)
  Week 17 | 55.75 (1.35) | 55.48 (1.40) | 49.45 (1.30) | 49.77 (1.30)
Statistical Analysis 1: Comparison: Survivors- SMSH Alone vs Survivors- SMSH+ TIPC; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at week 13 in linear mixed effects model; p = .45, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome was adjusted for in the model; Mean Difference (Final Values) = -1.41, 95% CI 2-sided [-5.22 to 2.39], Standard Error of Mean 1.94 — Mean of SMSH minus SMSH+TIPC
Statistical Analysis 2: Comparison: Survivors- SMSH Alone vs Survivors- SMSH+ TIPC; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at week 17 in linear mixed effects model; p = .82, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome was adjusted for in the model; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [-3.59 to 4.12], Standard Error of Mean 1.97 — Mean of SMSH minus SMSH+TIPC
Statistical Analysis 3: Comparison: Caregivers- SMSH Alone vs Caregivers- SMSH+ TIPC; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at week 13 in linear mixed effects model; p = .77, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome was adjusted for in the model; Mean Difference (Final Values) = 0.55, 95% CI 2-sided [-3.13 to 4.23], Standard Error of Mean 1.88 — Mean of SMSH minus SMSH+TIPC
Statistical Analysis 4: Comparison: Caregivers- SMSH Alone vs Caregivers- SMSH+ TIPC; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at week 17 in linear mixed effects model; p = .86, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome was adjusted for in the model; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-3.98 to 3.34], Standard Error of Mean 1.87 — Mean of SMSH minus SMSH+TIPC

ADVERSE EVENTS:
Time Frame: Each participant was assessed for adverse events at baseline (week 0), weekly for 12 weeks, and then at weeks 13 and 17 follow-ups or up until their attrition date if applicable.
Description: Adverse events/serious adverse events were identified during the implementation of the experimental protocols and were monitored by the Investigators in several ways: 1) Interviewers could identify both serious adverse events and/or adverse events during the completion of telephone interviews or telephone calls to schedule telephone interviews; 2) The interventionists could identify both serious adverse events and/or adverse events during their telephone contacts with the participants.
Groups:
- Survivors- SMSH Alone for 4 Weeks, Depression/Anxiety Responders Continued With SMSH Alone Week 5-12; Caregivers-SMSH Alone for 4 Weeks, Depression/Anxiety Responders Continued: The Symptom Management and Survivorship Handbook is a self-care management handbook with each symptom chapter presented in an identical format: what the symptom is, how people describe the symptom, the causes of the symptom, strategies for managing the symptom and resources. The Handbook was available in English and Spanish. Each weekly call began with a symptom assessment. For each symptom rated at 4 or higher on a 0-10 scale of severity, survivors and caregivers were referred for symptom self-management. After 4 weeks, depression or anxiety responders in the SMSH alone group continued with the SMSH alone for weeks 5-12. Depression or anxiety responders are survivors who started at severe at onset and ended at moderate or mild at a given time point (e.g., week 4), and survivors who started at moderate and ended at mild. At week 13, the survivor and caregiver were each called to complete the second assessment and at week 17 they were called to complete the third and final assessment.
Arm/Group | Survivors- SMSH Alone for 4 Weeks, Depression/Anxiety Responders Continued With SMSH Alone Week 5-12 | Survivors-SMSH Alone for 4 Weeks, Depression/Anxiety Non-responders Continued SMSH Alone Weeks 5-12 | Survivors- SMSH Alone for 4 Weeks, Depression/Anxiety Non-responders Continued SMSH+TIPC Weeks 5-12 | Survivors SMSH+TIPC During Weeks 1-8 Followed by SMSH Alone During Weeks 9-12 | Caregivers-SMSH Alone for 4 Weeks, Depression/Anxiety Responders Continued | Caregivers-SMSH Alone for 4 Weeks, Depression/Anxiety Non-responders Continued SMSH Alone Weeks 5-12 | Caregivers- SMSH Alone for 4 Weeks, Depression/Anxiety Non-responders Continued SMSH+TIPC Weeks 5-12 | Caregivers SMSH+TIPC During Weeks 1-8 Followed by SMSH Alone During Weeks 9-12 | Survivor Drop-outs From SMSH Alone Prior to Week 4 | Caregiver Drop-outs From SMSH Alone Prior to Week 4
All-Cause Mortality (participants affected / at risk) | 5/166 | 3/44 | 1/44 | 4/97 | 0/166 | 0/44 | 0/44 | 0/97 | 1/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/166 | 0/44 | 0/44 | 0/97 | 0/166 | 0/44 | 0/44 | 0/97 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/166 | 0/44 | 0/44 | 0/97 | 0/166 | 0/44 | 0/44 | 0/97 | 0/23 | 0/23

LIMITATIONS AND CAVEATS:
The larger than planned number of survivor-caregiver dyads with survivors responding to SMSH alone resulted in larger than planned number of participants in the first randomization and smaller number in the second randomization. There was a larger than planned number of responders to SMSH alone after 4 weeks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT03743415/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/15/NCT03743415/ICF_000.pdf